CLINICAL TRIAL: NCT01220765
Title: Assessment of Capnography in Monitoring Patients During Nurse Administered Deep Sedation With Propofol
Brief Title: Capnography During Nurse Administered Propofol Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: CASA, Leiden (Unknown)
Responsible Party: drs. K. van Loon, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL 29266.041.09
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Alveolar Hypoventilation Resulting in Hypoxemia
Keywords: hypoxemia; capnography; sedation
MeSH Terms: conditions — Hypoxia | interventions — Capnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Patients randomized to the standard care group receive standard of care using pulse oximetry
- Capnography (Experimental): In the intervention group capnography is measured using a cannula under the nose connected to the capnograph. The capnographic device displays respiratory rate, end-tidal carbon dioxide (ETCO2) levels, and continuous waveforms.
  Interventions: Device: Capnography

INTERVENTIONS:
Device: Capnography — In the capnography arm, respiratory monitoring is performed with pulse oximetry and capnography. If the capnogram indicates sub-optimal ventilation and/or apnea, denoted as a flat line on the capnometer for ≥ 15 seconds, a respiratory rate ≤ 6, or a end-tidal CO2 > 50 mmHg, medical staff will intervene by arousing the patient, performing chinlift or jawthrust, abandon from giving additional propofol, or provision of oxygen. The nurse qualified in sedation management will assess capnography him/ herself.
  Other Names: Capnograph, Capnostream TM 20, Oridion Medical 1987 ltd.
  Arms: Capnography

SUMMARY:
Rationale: The current standard of respiratory monitoring for patients during deep sedation is continuous pulse oximetry with visual assessment of the patient. Clinical research has demonstrated that depressed respiratory activity is a principal risk factor for hypoxemia during sedation. Capnography may provide early detection of alveolar hypoventilation before hypoxemia has occurred in nonintubated patients and thereby improve patient safety during sedation.

Objective: At the Centre for Contraception, Sexuality and Abortion Leiden, abortion procedures are performed under deep sedation using propofol. Patient's monitoring is performed by nurses qualified in patient sedation management, using pulse oximetry and their clinical judgement. The aim of this study is to examine the effectiveness of capnography in early detection of alveolar hypoventilation during deep sedation in comparison to standard monitoring with pulse oximetry in abortion procedures.

Study design: This protocol describes a prospective, open, randomized controlled trial with two study arms. All patients receive standard care of monitoring performed by the medical staff. The study investigates whether capnography prevents patients from having respiratory events during deep sedation in abortion procedures by early detection and therapy. Patients randomized to the standard care group receive standard of respiratory monitoring using pulse oximetry. In the capnography arm, respiratory monitoring is performed with pulse oximetry and capnography.

Study population: The study population comprises female patients (≥ 18 years) undergoing abortion procedures during first or second trimester pregnancies. Abortion procedures are performed until 22 weeks of gestational age.

Capnography: In addition application of capnography during deep sedation with propofol is performed. Before the trial starts, all nurses qualified in patient sedation management and abortion doctors will be trained in assessment of capnography. In the capnography arm, patients' breathing is additionally monitored with capnography. If alveolar hypoventilation is detected medical staff will intervene by arousing the patient, performing chin lift, repositioning the head, provision of oxygen, or abandon from giving additional propofol. These interventions represent the standard of care currently used by the clinical staff to respond to hypoventilation and hypoxemia.

Main study parameters/endpoints: The primary outcome is the occurrence of oxygen saturations to ≤90% in the population, as measured by continuous pulse oximetry. Secondary study outcomes include occurrence of oxygen saturations < 80%, dose of administered propofol, arousal or movement of the patient during the procedure, airway interventions, early termination of the procedure due to respiratory problems, episodes of bradycardia, and administration of atropine.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks related to the conduct of this study are negligible and the burden minimal. Patients in both groups receive the current standard of care. Patients randomized in the capnography group could get benefit from the addition of capnography to the monitoring by early detection of alveolar hypoventilation. Capnography is a noninvasive measurement by means of a cannula under the nose, which before the sedation may tickle, but during sedation no inconvenience is expected.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Since sedation is increasingly administered by non-anesthesiologists, patient safety during sedation became of increased interest by the Joint Commission for Accreditation of Healthcare Organisations (JCAHO). The current standard of respiratory monitoring for patients during sedation is continuous pulse oximetry with visual assessment of the patient. Clinical research has demonstrated that hypoxemia, secondary to depressed respiratory activity, is a principal risk during sedation. Microstream capnography is a relatively new technology for carbon dioxide (CO2) monitoring. The technique is based on emission of selective infrared wavelengths exactly matching for CO2 absorption. Due to this efficient and selective emission process only small samples of CO2 are necessary to detect alveolar hypoventilation, and accuracy is maintained with a low flow sample rate. Therefore, capnography can provide more useful information on the frequency, effectiveness and regularity of ventilation, than pulse oximetry during procedures accomplished under deep sedation. According to previous reports capnography provides early detection of alveolar hypoventilation before hypoxemia has occurred in nonintubated patients and thereby can improve patient safety during sedation.

   This study will provide new information on the efficacy of capnography for early detection of hypoxemia during nurse-administered propofol sedation in adults. Previous studies, involving a paediatric randomized study and a study in adult gastrointestinal endoscopy, were outcome studies with capnography in patients sedated with midazolam in combination with fentanyl or meperidine.4 5 Therefore, we will assess the efficacy of interventions based on capnographic monitoring of respiratory function in nurse-administered propofol sedation. In previously conducted studies independent observers monitored the capnographic display and prompted the medical team of the changes in respiratory activity. In the following clinical trial we will examine normal practice by assessment of the capnogram by the nurse qualified in sedation management.
2. OBJECTIVES At the Centre for Contraception, Sexuality and Abortion (CASA) Leiden abortion procedures are performed under deep sedation using propofol. These procedures are not attended by an anesthesiologist and patient's monitoring is performed by nurses qualified in patient sedation management, using pulse oximetry and their clinical judgement. Supplementary oxygen is not routinely given.

   The purpose of this study is to investigate the use of capnography to improve patient safety during deep sedation. This study examines the effectiveness of capnography in early detection and therapy of alveolar hypoventilation during deep sedation in comparison to standard monitoring with pulse oximetry in abortion procedures. The randomized controlled trial determines whether utilizing capnography in women undergoing deep sedation with propofol (monotherapy) for abortion procedures will provide early detection of suboptimal ventilation and reduce hypoxemia. Unlike previous studies we are determined to investigate daily practice when nurses qualified in sedation management assess capnography instead of an independent observer assessing capnography. Therefore, all nurses qualified in patient sedation management and abortion doctors will be trained in assessment of capnography before the trial starts.

   The implications of this study for monitoring deep sedation may be generalized to all healthy patients having minimal invasive procedures, particularly when a trained anesthesiologist is not in attendance.
3. STUDY DESIGN This protocol describes a prospective, open, randomized controlled trial with two study arms. All patients receive standard care of monitoring performed by the medical staff. The study examines whether capnography prevents patients from having respiratory events during deep sedation in abortion procedures.Patients randomized to the standard care group receive standard of care using pulse oximetry. In the capnography arm, respiratory monitoring is performed with pulse oximetry and capnography. If the capnogram indicates sub-optimal ventilation and/or apnea, denoted as a flat line on the capnometer for ≥ 15 seconds, a respiratory rate ≤ 6, or a end-tidal CO2 > 50 mmHg, medical staff will intervene by arousing the patient, performing chinlift or jawthrust, abandon from giving additional propofol, or provision of oxygen. The nurse qualified in sedation management will assess capnography him/ herself. Medical staff and patients are not blinded for the allocation assignment and the study has an open design.
4. STUDY POPULATION 4.1 Population Participants are recruited at the Centre for Contraception, Sexuality and Abortion Leiden, the Netherlands. The study population comprises female patients (≥ 18 years) undergoing abortion procedures during first or second trimester pregnancies.

   4.2 Inclusion criteria Patients were considered for enrolment if they fulfil all of the following inclusion criteria: age 18 years or older, abortion procedures performed until 22 weeks of gestational age, American Society of Anaesthesiologists (ASA) classes I to II, and ability (mental competence) to give informed consent.

   4.3 Exclusion criteria Exclusion criteria were inability to provide informed consent, history of allergic reactions to propofol, soybeans or egg proteins, American Society of Anaesthesiologists (ASA) classes III- V, sleep apnea syndrome, and seizure disorders.

   4.4 Sample size calculation The sample size calculation for the prospective randomized controlled trial is based on a comparison of two proportions. The proportion of patients developing hypoxemia during sedation is reported between 47% and 51% in observational studies.1 2 Qadeer et al. reported a reduction of hypoxemia (saturation <90%) with additional capnography monitoring from 69% to 46% and Lightdale et al. reported a reduction of hypoxemia (saturation <95%) in children from 24% to 11%.4 5 Based on an observation of daily practice in 58 patients at the CASA clinic Leiden hypoxemia (oxygen saturation < 90%) was recorded in 12 patients, corresponding to an incidence of 20.7%. To show a decrease in hypoxemia from 20% to 10% with a significance level of 0.05 and a power of 0.80, 219 patients are required within each arm, yielding 440 patients to be included in total. Give the annual number of 1600 patients and expecting a participation rate of 60%, we expect to include these patients within a period of 24 weeks.
5. METHODS 5.1 Study parameters/endpoints

5.1.1 Main study parameter/ endpoint The primary outcome is the occurrence of oxygen saturations to <90% in the population, measured by continuous pulse oximetry.

5.1.2 Secondary study parameters/endpoints Secondary study outcomes include occurrence of oxygen saturations to <80%, total administered propofol dose, airway interventions (repositioning the head, chinlift, supplemental oxygen, bag-mask ventilation), problems during the abortion procedure (e.g. arousal or movement of the patient), early termination of the procedure due to respiratory problems, episodes of bradycardia, administration of atropine.

5.1.3 Other study parameters Carbon dioxide monitoring with capnography will provide the following parameters: apnea (absence of respiratory activity) denoted as a flat line on the capnometer for ≥ 15 seconds, abnormal ventilation denoted as a respiratory rate ≤ 6, and end-tidal CO2 > 50 mmHg (CO2 > 6.7 kPa).

Baseline values are age, height, body weight, duration of pregnancy, American Society of Anaesthesiologists class, smoking, abuse of alcohol or drugs, and use of soporifics.

5.2 Randomisation, blinding and treatment allocation During the trial patients are randomly assigned to the capnography group (standard care and monitoring with capnography) or the control group (standard care) by randomisation. The randomisation is computer-generated and stratified for each abortion doctor.

Participants are recruited by an independent observer or nurse. The patient and medical staff will not be blinded to the allocation assignment and also the independent observer is aware of the randomisation assignment before the start of the procedure.

5.3 Study procedures

* Daily practice at the CASA clinic: If patients opt for an abortion procedure after five days of statutory reflection they are coming to the clinic with an appointment. Before any procedure starts, patients have again a conversation with a doctor or nurse about their decision to have an abortion. If an abortion is inevitable and pregnancy lasts no longer than 16 weeks, the patient is immediately admitted to the clinic. If an abortion is inevitable and pregnancy lasts between 16 and 22 weeks, cervical priming with misoprostol is administered at least 90 minutes before the abortion procedure.
* A routinely performed health questionnaire, blood pressure, heart rate and blood group determination are performed in preparation for the procedure. Peripheral venous access is established at the holding area. Baseline characteristics for the study are obtained by this routinely performed questionnaire including health questions (e.g. weight, height, and smoking).
* Patients are asked to be a participant for this study by one of the nurses or by the researcher at the holding area. They receive an information letter and are able to question the researcher about their participation.
* Before the procedure starts monitoring, including pulse oximetry and blood pressure, is attached to each patient
* All patients receive standard monitoring with continuous display of pulse oximetry and heart rate. In the intervention group capnography is measured using a cannula under the nose connected to the capnograph, Capnostream TM 20, Oridion Medical 1987 ltd. This capnographic device displays respiratory rate, end-tidal carbon dioxide (ETCO2) levels, and continuous waveforms.
* All patients are sedated with an initial dose of 100 milligrams (mg) propofol. In addition 20-50 mg propofol is administered when patient discomfort or lighter levels of sedation are noticed. The nurse qualified in sedation management determines the doses of propofol on a previously described sedation protocol for the CASA clinics. Local anesthesia of the cervix is performed with 10-20 ml lidocaine 1%.
* When the abortion procedure has finished patients are monitored at the recovery area. If they are fully awake and no extensive bleeding has occurred, they are allowed to leave the clinic.

5.4 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. It should however be noted that patients during sedation no longer have the ability to express their wishes.

ELIGIBILITY:
Inclusion Criteria:

* Patients were considered for enrolment if they fulfil all of the following inclusion criteria: age 18 years or older, abortion procedures performed until 22 weeks of gestational age, American Society of Anaesthesiologists (ASA) classes I to II, and ability (mental competence) to give informed consent.

Exclusion Criteria:

* Exclusion criteria were inability to provide informed consent, history of allergic reactions to propofol, soybeans or egg proteins, American Society of Anaesthesiologists (ASA) classes III- V, sleep apnea syndrome, and seizure disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having saturations (SpO2 below 90%) in the two arms | Desaturations during the sedation procedure, within 1 hour after administering the first propofol dose
  Occurrence of oxygen saturations below 90% measured by continuous pulse oximetry in the two study arms; capnography vs. standard care

SECONDARY OUTCOMES:
proportion of patients necessitating airway interventions | Airway interventions during the sedation procedure within 1 hour after the first propofol dose
  Secondary study outcomes include airway interventions (repositioning the head, chinlift, supplemental oxygen, bag-mask ventilation), problems during the abortion procedure (e.g. arousal or movement of the patient), early termination of the procedure due to respiratory problems, episodes of bradycardia, administration of atropine.
Proportion of patients having deep desaturations (SpO2 below 80%) in the two study arms | Desaturations during the sedation procedure, within 1 hour after the first propofol dose
  Occurrence of oxygen saturations below 80% measured by continuous pulse oximetry in the two study arms; capnography vs. standard care

CONTACTS AND LOCATIONS:
Locations (1):
- CASA, Centre for Contraception, Sexuality and Abortion clinic,, Leiden, Netherlands

REFERENCES:
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Shermock KM, Morrow JB, Conwell DL, Trolli PA, Maurer WG. Gastroenterologist-administered propofol versus meperidine and midazolam for advanced upper endoscopy: a prospective, randomized trial. Gastroenterology. 2002 Jul;123(1):8-16. doi: 10.1053/gast.2002.34232. PMID 12105827
- [Background] Griffin SM, Chung SC, Leung JW, Li AK. Effect of intranasal oxygen on hypoxia and tachycardia during endoscopic cholangiopancreatography. BMJ. 1990 Jan 13;300(6717):83-4. doi: 10.1136/bmj.300.6717.83. No abstract available. PMID 2105779
- [Background] Colman Y, Krauss B. Microstream capnograpy technology: a new approach to an old problem. J Clin Monit Comput. 1999 Aug;15(6):403-9. doi: 10.1023/a:1009981115299. PMID 12578035
- [Background] Lightdale JR, Goldmann DA, Feldman HA, Newburg AR, DiNardo JA, Fox VL. Microstream capnography improves patient monitoring during moderate sedation: a randomized, controlled trial. Pediatrics. 2006 Jun;117(6):e1170-8. doi: 10.1542/peds.2005-1709. Epub 2006 May 15. PMID 16702250
- [Background] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079
- [Background] Grobbee DE, Hoes AW. Randomized trials. In: Grobbee DE, Hoes AW, editors. Clinical Epidemiology. Sudbury: Jones and Bartlett; 2008. p. 270-287.
- [Background] Clarke JP. Sedation for endoscopy: the safe use of propofol by general practitioners. Med J Aust. 2002 Aug 5;177(3):163-4; author reply 165. doi: 10.5694/j.1326-5377.2002.tb04712.x. No abstract available. PMID 12149092